CLINICAL TRIAL: NCT04830527
Title: Development and Evaluation of an Ecological Momentary Assessment (EMA) Baseline Screening System for Therapists Who Treat Youths With Depressive Symptoms
Brief Title: EMA Baseline Screening System for Therapists Who Treat Youths With Depressive Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to the difficulty in recruiting cases during a pandemic period.
Sponsor: Vania Martínez-Nahuel (Other)
Collaborators: ANID - Millennium Science Initiative Program - NCS17_03 Millennium Nucleus to Improve the Mental Health of Adolescents and Youths (Imhay), Santiago, Chile (Unknown); Millennium Institute on Immunology and Immunotherapy (Other); Center for Psychotherapy Research, University Hospital Heidelberg, Heidelberg, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Vania Martínez-Nahuel, Dr., University of Chile
Organization: University of Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 030-2020
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Depressive Symptoms
Keywords: depression; therapeutic alliance; youth; Ecological Momentary Assessment; e-mental Health; e-Health; adherence
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in experimental group will receive EMA prompts. Therapists in this group will receive a summarized PDF report before the beginning of the first psychotherapy session. The report will include graphic summarized data from the EMA prompts.
  Interventions: Behavioral: EMA prompting for patients; Behavioral: PDF Reports for therapists
- Control group (Active Comparator): Patients in control group will receive the EMA prompts in the same manner as patients in the experimental group.
  Therapists in this group will not receive the PDF reports, and instead will get raw scores from a screening evaluation conducted with patients in the recruitment phase of the study.
  Interventions: Behavioral: EMA prompting for patients

INTERVENTIONS:
Behavioral: EMA prompting for patients — EMA prompting will consist of the delivery of the PHQ-4 and PANAS questionnaires, as well as basic identification, therapy motivations and expectations, location, current activity and social interactions.
  These prompts will be presented to patients during a 7 day period, 5 times per day.
Behavioral: PDF Reports for therapists — After the patients' EMA data is collected, a previously designed R script will summarize and transform the data into a brief and graphic report for therapists in the experimental arm of the study. These reports are intended to provide detailed information about the patients' mood, anxiety levels, positive and negative affects, as well as crossed data such as mood according to location, anxiety according to activity, etc.
  Arms: Intervention group

SUMMARY:
Youth depression is a matter of concern worldwide. It affects an important part of the young population around the world and its consequences both physically and mentally make this issue an important research field for psychologists and other health related professionals (Zuckerbrot, Cheung, Jensen, Stein & Laraque, 2018). Two of the biggest challenges that clinicians and researchers face when dealing with youth depression are adherence and the establishment of a therapeutic alliance (TA; Nock & Ferriter, 2005). While several treatments are available to relief depressive symptomatology in youths, a significant number do not access them for a variety of reasons (DiMatteo, Lepper & Corgan, 2000). In the last decades, substantial research has been conducted on how youths and the general population perceive therapy, and different methods have been developed to assess clients and therapists in order to improve outcomes and other aspects of the psychotherapy process, such as feedback tools and real-time measurements like Ecological Momentary Assessment (EMA) (Shiffman, et al., 2008). With the aid of Information Communication Technologies (ICTs) and eMental Health strategies, feedback and assessment tools can be presented in a friendly manner, providing a novel way to possibly improving adherence rates and TA scores. This study aims to develop and test the effectiveness of an Ecological Momentary Assessment mobile application to improve initial adherence and TA in psychotherapy for youths with depression.

The hypotheses for this trial are:

1. Applying an EMA baseline screening application one week before the beginning of treatment for youth depression will significantly improve the TA.
2. Applying an EMA baseline screening application one week before the beginning of treatment for youth depression will significantly improve initial adherence.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Owning a mobile phone with permanent access to the internet,
* Scoring from eleven to nineteen points in the PHQ-9 questionnaire.
* Having completed the eighth grade of basic education.

Exclusion Criteria for Patients:

* Being diagnosed with Depression with psychotic symptoms,
* Having a depressive episode as part of a bipolar disorder diagnosis
* Having suicidal thoughts and/or behaviour as measured by the PHQ-9 and evaluated by the physician.
* Alcohol and/or substance abuse.

Inclusion Criteria for Therapists:

- Having 1 or more years of clinical experience.

Exclusion Criteria for Therapists:

* Having less than 1 year of clinical experience.
* Having participated in the design of PDF reports.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Working Alliance Inventory, Patient Form (WAI-P) | Immediately after the end of first three psychotherapy sessions.
  Likert scale with answers that range from 1 to 7. Higher scores suggest a better perception of the Therapeutic Alliance.

SECONDARY OUTCOMES:
Working Alliance Inventory, Therapist Form (WAI-T) | Immediately after the end of first three psychotherapy sessions.
  Likert scale with answers that range from 1 to 7. Higher scores suggest a better perception of the Therapeutic Alliance.
Assistance to sessions | Immediately after the end of first three psychotherapy sessions.
  Assistance to sessions will be registered by therapists as a measurement of initial adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- CEMERA, Faculty of Medicine, Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abras, C., Maloney-Krichmar, D., Preece, J. (2004) User-Centered Design. In Bainbridge, W. Encyclopedia of Human-Computer Interaction. Thousand Oaks: Sage Publications.
- [Background] Borghero F, Martinez V, Zitko P, Vohringer PA, Cavada G, Rojas G. [Screening depressive episodes in adolescents. Validation of the Patient Health Questionnaire-9 (PHQ-9)]. Rev Med Chil. 2018 Apr;146(4):479-486. doi: 10.4067/s0034-98872018000400479. Spanish. PMID 29999123
- [Background] Cipriani A, Zhou X, Del Giovane C, Hetrick SE, Qin B, Whittington C, Coghill D, Zhang Y, Hazell P, Leucht S, Cuijpers P, Pu J, Cohen D, Ravindran AV, Liu Y, Michael KD, Yang L, Liu L, Xie P. Comparative efficacy and tolerability of antidepressants for major depressive disorder in children and adolescents: a network meta-analysis. Lancet. 2016 Aug 27;388(10047):881-90. doi: 10.1016/S0140-6736(16)30385-3. Epub 2016 Jun 8. PMID 27289172
- [Background] Clark MS, Jansen KL, Cloy JA. Treatment of childhood and adolescent depression. Am Fam Physician. 2012 Sep 1;86(5):442-8. PMID 22963063
- [Background] Cox GR, Callahan P, Churchill R, Hunot V, Merry SN, Parker AG, Hetrick SE. Psychological therapies versus antidepressant medication, alone and in combination for depression in children and adolescents. Cochrane Database Syst Rev. 2014 Nov 30;2014(11):CD008324. doi: 10.1002/14651858.CD008324.pub3. PMID 25433518
- [Background] David-Ferdon C, Kaslow NJ. Evidence-based psychosocial treatments for child and adolescent depression. J Clin Child Adolesc Psychol. 2008 Jan;37(1):62-104. doi: 10.1080/15374410701817865. PMID 18444054
- [Background] Eapen V, Crncec R. Strategies and challenges in the management of adolescent depression. Curr Opin Psychiatry. 2012 Jan;25(1):7-13. doi: 10.1097/YCO.0b013e32834de3bd. PMID 22156932
- [Background] Fernández, O., Pérez, C., Gloger, S., Krause, M., (2015) Importancia de los cambios iniciales en psicoterapia con jovenes, Terapia Psicológica, (33)3, pp. 247 - 255.
- [Background] Fernández, O. M., Herrera-Salinas, P. & Escobar-Martínez, M. J. (2016). youthes en Psicoterapia: Su Representación de la Relación Terapéutica. Revista Latinoamericana de Ciencias Sociales, Niñez y Juventud, 14 (1), pp. 559-575.
- [Background] Fernandez, O.M., Krause, M., & Pérez, J.C. (2016). Therapeutic alliance in the initial phase of psychotherapy with ado- lescents: different perspectives and their association with therapeutic outcomes. Research in Psychotherapy: Psychopathology, Process and Outcome, 19(1), 1-9. doi: 10.4081/ripppo.2016.180
- [Background] Goodyer IM, Reynolds S, Barrett B, Byford S, Dubicka B, Hill J, Holland F, Kelvin R, Midgley N, Roberts C, Senior R, Target M, Widmer B, Wilkinson P, Fonagy P. Cognitive-behavioural therapy and short-term psychoanalytic psychotherapy versus brief psychosocial intervention in adolescents with unipolar major depression (IMPACT): a multicentre, pragmatic, observer-blind, randomised controlled trial. Health Technol Assess. 2017 Mar;21(12):1-94. doi: 10.3310/hta21120. PMID 28394249
- [Background] Hatcher, R., & Gillaspy, J., (2006) Development and validation of a revised short version of the working alliance inventory, Psychotherapy Research, 16:1, 12-25, DOI: 10.1080/10503300500352500
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kelders SM, Kok RN, Ossebaard HC, Van Gemert-Pijnen JE. Persuasive system design does matter: a systematic review of adherence to web-based interventions. J Med Internet Res. 2012 Nov 14;14(6):e152. doi: 10.2196/jmir.2104. PMID 23151820
- [Background] Lal S, Adair CE. E-mental health: a rapid review of the literature. Psychiatr Serv. 2014 Jan 1;65(1):24-32. doi: 10.1176/appi.ps.201300009. PMID 24081188
- [Background] Lambert MJ, Whipple JL, Smart DW, Vermeersch DA, Nielsen SL, Hawkins EJ. The effects of providing therapists with feedback on patient progress during psychotherapy: are outcomes enhanced? Psychother Res. 2001 Mar;11(1):49-68. doi: 10.1080/713663852. PMID 25849877
- [Background] Lambert MJ. Maximizing Psychotherapy Outcome beyond Evidence-Based Medicine. Psychother Psychosom. 2017;86(2):80-89. doi: 10.1159/000455170. Epub 2017 Feb 10. PMID 28183083
- [Background] Luciano JV, Bertsch J, Salvador-Carulla L, Tomas JM, Fernandez A, Pinto-Meza A, Haro JM, Palao DJ, Serrano-Blanco A. Factor structure, internal consistency and construct validity of the Sheehan Disability Scale in a Spanish primary care sample. J Eval Clin Pract. 2010 Oct;16(5):895-901. doi: 10.1111/j.1365-2753.2009.01211.x. PMID 20626541
- [Background] Lewinsohn PM, Clarke GN. Psychosocial treatments for adolescent depression. Clin Psychol Rev. 1999 Apr;19(3):329-42. doi: 10.1016/s0272-7358(98)00055-5. PMID 10097874
- [Background] Michael KD, Crowley SL. How effective are treatments for child and adolescent depression? A meta-analytic review. Clin Psychol Rev. 2002 Mar;22(2):247-69. doi: 10.1016/s0272-7358(01)00089-7. PMID 11806021
- [Background] Nock MK, Ferriter C. Parent management of attendance and adherence in child and adolescent therapy: a conceptual and empirical review. Clin Child Fam Psychol Rev. 2005 Jun;8(2):149-66. doi: 10.1007/s10567-005-4753-0. PMID 15984084
- [Background] O'Dea B, Calear AL, Perry Y. Is e-health the answer to gaps in adolescent mental health service provision? Curr Opin Psychiatry. 2015 Jul;28(4):336-42. doi: 10.1097/YCO.0000000000000170. PMID 26001926
- [Background] Pacheco, B. & Aránguiz, C., (2011) Factores relacionados a la adherencia a tratamiento en youthes con depresión, Revista Chilena de Neuro-Psiquiatría, 49(1), pp. 69-78.
- [Background] Riper H, Andersson G, Christensen H, Cuijpers P, Lange A, Eysenbach G. Theme issue on e-mental health: a growing field in internet research. J Med Internet Res. 2010 Dec 19;12(5):e74. doi: 10.2196/jmir.1713. PMID 21169177
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Shimokawa K, Lambert MJ, Smart DW. Enhancing treatment outcome of patients at risk of treatment failure: meta-analytic and mega-analytic review of a psychotherapy quality assurance system. J Consult Clin Psychol. 2010 Jun;78(3):298-311. doi: 10.1037/a0019247. PMID 20515206
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Shirk SR, Karver M. Prediction of treatment outcome from relationship variables in child and adolescent therapy: a meta-analytic review. J Consult Clin Psychol. 2003 Jun;71(3):452-64. doi: 10.1037/0022-006x.71.3.452. PMID 12795570
- [Background] Silk JS, Forbes EE, Whalen DJ, Jakubcak JL, Thompson WK, Ryan ND, Axelson DA, Birmaher B, Dahl RE. Daily emotional dynamics in depressed youth: a cell phone ecological momentary assessment study. J Exp Child Psychol. 2011 Oct;110(2):241-57. doi: 10.1016/j.jecp.2010.10.007. Epub 2010 Nov 26. PMID 21112595
- [Background] Weersing VR, Brent DA, Rozenman MS, Gonzalez A, Jeffreys M, Dickerson JF, Lynch FL, Porta G, Iyengar S. Brief Behavioral Therapy for Pediatric Anxiety and Depression in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jun 1;74(6):571-578. doi: 10.1001/jamapsychiatry.2017.0429. PMID 28423145
- [Background] Weisz JR, Kuppens S, Ng MY, Eckshtain D, Ugueto AM, Vaughn-Coaxum R, Jensen-Doss A, Hawley KM, Krumholz Marchette LS, Chu BC, Weersing VR, Fordwood SR. What five decades of research tells us about the effects of youth psychological therapy: A multilevel meta-analysis and implications for science and practice. Am Psychol. 2017 Feb-Mar;72(2):79-117. doi: 10.1037/a0040360. PMID 28221063